CLINICAL TRIAL: NCT00630747
Title: An Open-Label Extension of Study TKT024 Evaluating Long-Term Safety and Clinical Outcomes in MPS II Patients Receiving Iduronate-2-Sulfatase Enzyme Replacement Therapy
Brief Title: Extension of Study TKT024 Evaluating Long-Term Safety and Clinical Outcomes in MPS II Patients Receiving Idursulfase
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TKT024EXT; 2004-002743-27 (EudraCT Number)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Hunter Syndrome; Mucopolysaccharidosis II (MPS II)
Keywords: Hunter syndrome; hunters syndrome; hunter's syndrome; hunter disease; hunters disease; hunter's disease; MPS II; MPSII; MPS2; MPS 2; mucopolysaccharides; lysosomal storage disease; lysosomal storage disorder; chronic ear infection; enlarged adenoids; mps symptoms; mps diagnosis; mps ii therapy; MPS II treatment; ert treatment; elaprase; idursulfase; iduronate sulfatase; iduronate 2 sulfatase; enzyme replacement therapy; hunter syndrome treatment; hunter's syndrome treatment; hunter syndrome therapy; hunter's disease treatment; mps society
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death; Lysosomal Storage Diseases | interventions — idursulfase; Iduronate Sulfatase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Idursulfase (Experimental)
  Interventions: Biological: Idursulfase

INTERVENTIONS:
Biological: Idursulfase — Solution for intravenous infusion, 0.5 mg/kg once-weekly
  Other Names: Elaprase®; iduronate-2-sulfatase

SUMMARY:
Study TKT024EXT was a long-term, single-arm, open-label extension of Study TKT024, a one year Phase 2/Phase 3 registration study. The primary objective of this extension study was to collect long-term safety and clinical outcome data in Mucopolysaccharidosis II (MPS II), also known as Hunter Syndrome, from the Phase 2/Phase 3 Study TKT024. All patients enrolling into this study received weekly active treatment with idursulfase, the primary dosing regimen investigated in Study TKT024.

Hunter Syndrome is an X-linked recessive lysosomal storage disease caused by a deficiency of iduronate-2-sulfatase, an enzyme required to catabolize glycosaminoglycans (GAGS) in cells. As a result, GAGs accumulate in the lysosomes leading to cellular engorgement, organomegaly, tissue destruction, and organ system dysfunction. Hunter Syndrome is a rare disease with an estimated incidence of 1 in 162,000 live births.

DETAILED DESCRIPTION:
Study TKT024EXT was conducted in 2 phases. The first phase ("Phase I") was 2 years (104 weeks) in duration and consisted of weekly infusions of IV idursulfase (0.5 mg/kg), and the collection of patients' safety and clinical outcomes. Week 105 defined the beginning of the second phase of the study. The second phase ("Phase II") consisted of weekly infusions of IV idursulfase (0.5 mg/kg) and the monitoring of patients for safety (via collection of adverse events, concomitant medications, and vital signs). Study completion was defined as the time a patient either transitioned to commercially available idursulfase or discontinued this study.

Idursulfase was administered to patients as a continuous IV infusion at a dose of 0.5 mg of protein per kg of body weight (0.5 mg/kg). Final evaluations from Study TKT024, the one-year predecessor Phase 2/Phase 3 registration study, served as the baseline assessments for the TKT024EXT study. Forced vital capacity (FVC) and the 6-minute walk test (6MWT) continued to be the primary clinical outcomes of TKT024EXT study. Efficacy outcomes were evaluated over the course of 2 years and were determined at 4-month intervals during the first year (ie, Weeks 18, 36, and 53) and at 6-month intervals in the second year (ie, Weeks 79 and 105). Safety outcomes were assessed throughout the duration of the study. The safety and clinical testing performed in the TKT024EXT study were identical to those performed in the double-blind phase of Study TKT024.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have completed the double-blind phase of Study TKT024, defined as completing the Week 53 final evaluations.
* Patient, patient's parent(s), or legally authorized representative must have voluntarily signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient.

Exclusion Criteria:

* Patient has received treatment with an investigational therapy other than iduronate-2-sulfatase in Study TKT024 within the past 60 days.
* Patient is unable to comply with the protocol (e.g., due to a medical condition such as cervical cord compression or uncooperative attitude) or is unlikely to complete the study, as determined by the investigator.
* Patient has experienced an adverse reaction to study drug in Study TKT024, which contraindicates further treatment with idursulfase.
* Patient with known hypersensitivity to any of the components of idursulfase.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2004-09-13 (Actual); Primary Completion 2008-01-31 (Actual); Study Completion 2008-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (52):
- United States (16):
  - St. Joseph's Hospital, Phoenix, Arizona
  - Pediatric Clinical Research Center, Children's Hospital Oakland, Oakland, California
  - The Children's Hospital, Denver, Colorado
  - Harbin Clinic, Rome, Georgia
  - Mid-Illinois Hematology and Oncology Associates, Normal, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Children's Hospital Boston, Boston, Massachusetts
  - Saint Louis University Cardinal Glennon Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Upstate Medical University, State University of New York (SUNY), Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine Texas Children's Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
- Brazil (8):
  - Fundacao Universidade de Ciencias da Saude de Alagoas Governador Lamenha Filho / UNCISAL, Maceió, Alagoas
  - Clinica Casa de Saude Sao Joao, Barreiras, Estado de Bahia
  - c-HUPES/UFBA, Salvador, Estado de Bahia
  - Hospital Universitario da Faculdade de Medicina da Universidade Federal de Mato Grosso do Sul, Campo Grande, Mato Grosso do Sul
  - Instituto de Puericultura e Pediatria Martagao Gesteira / Hospital Pediatrico, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Servico de Genetica Medica, Porto Alegre, Rio Grande do Sul
  - UNIFESP Instituto de Oncologia Pediatrica, São Paulo, São Paulo
  - Instituto da Crianca / Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
- Canada (2):
  - The Hospital for Sick Children Research Institute, Toronto, Ontario
  - University of Montreal / Hopital Ste-Justine, Montreal, Quebec
- France (3):
  - Hopital Edouard Herriot, Lyon
  - Hopital de Hautepierre, Strasbourg
  - Hospital Ducuing, Toulouse
- Germany (6):
  - Universitatsklinikum Aachen Kinderklinik, Aachen
  - Universitatsklinik Dusseldorf Kinderklinik, Düsseldorf
  - Justus-Liebig Universitat, Giessen
  - Universitatsklinikum Gottingen, Göttingen
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Children's University Hospital Mainz AG, Mainz
- Italy (4):
  - Universita Milano Bicocca / Ospedale S. Gerardo, Milan
  - Universita degli Studi di Napoli Federico II, Napoli
  - Universita di Padova, Padua
  - Ospedale S. S. Annunziata, Savigliano
- Spitalul Clinic de Copii, Cluj-Napoca, Cluj, Romania
- Spain (2):
  - Servicio de Pediatria, Linares, Jaen
  - University Hospital Germans Trias i Pujol, Badalona
- Sweden (2):
  - Drottning Silvias Barnsjukhus, Gothenberg
  - Karolinska University Hospital, Stockholm
- United Kingdom (8):
  - Royal Surrey County Hospital, Guildford, Surrey
  - Bath and NE Somerset Primary Care Trust, Bath
  - Addenbrooke's Hospital, Cambridge
  - Derbyshire Children's Hospital, Derby
  - Royal Hospital for Sick Children, Glasgow
  - Great Ormond Street Hospital for Sick Children, London
  - Royal Manchester Children's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle

REFERENCES:
- [Background] Muenzer J, Gucsavas-Calikoglu M, McCandless SE, Schuetz TJ, Kimura A. A phase I/II clinical trial of enzyme replacement therapy in mucopolysaccharidosis II (Hunter syndrome). Mol Genet Metab. 2007 Mar;90(3):329-37. doi: 10.1016/j.ymgme.2006.09.001. Epub 2006 Dec 20. PMID 17185020
- [Background] Muenzer J, Wraith JE, Beck M, Giugliani R, Harmatz P, Eng CM, Vellodi A, Martin R, Ramaswami U, Gucsavas-Calikoglu M, Vijayaraghavan S, Wendt S, Puga AC, Ulbrich B, Shinawi M, Cleary M, Piper D, Conway AM, Kimura A. A phase II/III clinical study of enzyme replacement therapy with idursulfase in mucopolysaccharidosis II (Hunter syndrome). Genet Med. 2006 Aug;8(8):465-73. doi: 10.1097/01.gim.0000232477.37660.fb. PMID 16912578
- [Result] Muenzer J, Beck M, Eng CM, Giugliani R, Harmatz P, Martin R, Ramaswami U, Vellodi A, Wraith JE, Cleary M, Gucsavas-Calikoglu M, Puga AC, Shinawi M, Ulbrich B, Vijayaraghavan S, Wendt S, Conway AM, Rossi A, Whiteman DA, Kimura A. Long-term, open-labeled extension study of idursulfase in the treatment of Hunter syndrome. Genet Med. 2011 Feb;13(2):95-101. doi: 10.1097/GIM.0b013e3181fea459. PMID 21150784
- [Derived] Beusterien KM, Yeung JE, Pang F, Brazier J. Development of the multi-attribute Adolescent Health Utility Measure (AHUM). Health Qual Life Outcomes. 2012 Aug 28;10:102. doi: 10.1186/1477-7525-10-102. PMID 22929184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study allows participants in double-blind phase of Study TKT024 (NCT00069641), a 1 year Phase 2/3 registration study, to continue long-term idursulfase therapy and to allow placebo participants in TKT024 to receive active idursulfase treatment. The first participant enrolled on 13 Sep 2004. The study was conducted at 52 sites in 17 countries.
Pre-assignment Details: Participants were screened for entry based on their known medical histories and previous participation in the TKT024 study. Participants had to have completed Week 53 final evaluations in the TKT024 study. Participants were not to have received any treatment with an investigational therapy other than idursulfase within 60 days of study entry.
Groups:
- Idursulfase (0.5 mg/kg, IV, Once-weekly): Idursulfase 0.5 milligram per kilogram (mg/kg) administered by intravenous (IV) infusion once-weekly.
Period: Overall Study
Arm/Group | Idursulfase (0.5 mg/kg, IV, Once-weekly)
Started | 94
Participants Treated in Phase I of Study | 94
Completed | 85
Not Completed | 9
Not completed — Death | 1
Not completed — Transferred to Study TKT031NPU | 7
Not completed — Returned to country of origin | 1

BASELINE CHARACTERISTICS:
Groups:
- Idursulfase (0.5 mg/kg, IV, Once-weekly): Idursulfase 0.5 mg/kg administered by IV infusion once-weekly.
Arm/Group | Idursulfase (0.5 mg/kg, IV, Once-weekly)
Number analyzed (Participants) | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 70
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.52 (6.634)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 78
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 40
  North America | 34
  South America | 20
Baseline Percent Predicted Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: percent predicted FVC] | 56.160 (14.897)
Baseline Distance Walked in the 6-minute Walk Test (6MWT) [Mean (Standard Deviation); unit: meters (m)] | 400.3 (100.25)
Baseline Passive Joint Range of Motion (JROM) [Mean (Standard Deviation); unit: percentage of JROM] — Global JROM (% normal range of motion) is the average of 11 ratios multiplied by 100. Ratios are Left/Right means of passive range of motion in Shoulder (Flexion/Extension, Abduction, Internal/External Rotation), Elbow (Flexion/Extension), Wrist (Flexion/Extension), Index Finger (Flexion/Extension [Combined MCP, PIP, DIP motion]), Hip (Flexion/Extension, Abduction, Internal/External Rotation), Knee (Flexion/Extension), and Ankle (Dorsiflexion) divided by the normal range (American Academy of Orthopedic Surgeons and American Medical Association).
  percentage of JROM | 67.44 (9.042)
Baseline Combined Liver and Spleen Volume [Mean (Standard Deviation); unit: cubic centimeters (cc)] | 1504.8 (417.21)
Baseline Normalized Urine Glycosaminoglycans (GAG) Levels [Mean (Standard Deviation); unit: microgram(mcg)GAG/mg creatinine] | 361.96 (136.132)
Baseline Cardiac Left Ventricular Mass Index (LVMI) [Mean (Standard Deviation); unit: gram per meter^2 (g/m^2)] | 97.64 (36.606)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Percent Predicted Forced Vital Capacity (FVC) at Week 105
Description: Determined by spirometry. The change is calculated as Week 105 minus baseline.
Time Frame: Baseline and at Week 105
Population: All participants for whom percent predicted FVC were recorded at baseline and at Week 105.
Measure: Mean (Standard Error); unit: percent predicted FVC
Arm/Group | Idursulfase (0.5 mg/kg, IV, Once-weekly)
Number analyzed (Participants) | 85
percent predicted FVC | -0.056 (1.059)

2. Secondary Outcome: Change From Baseline in Mean Passive Joint Range of Motion (JROM) at Week 105
Description: Change was calculated as Week 105 minus baseline. Global JROM (% normal range of motion) is the average of 11 ratios multiplied by 100. Ratios are Left/Right means of passive range of motion in Shoulder (Flexion/Extension, Abduction, Internal/External Rotation), Elbow (Flexion/Extension), Wrist (Flexion/Extension), Index Finger (Flexion/Extension [Combined Metacarpophalangeal joint (MCP), Proximal interphalangeal joint (PIP), Distal interphalangeal joint (DIP) motion]), Hip (Flexion/Extension, Abduction, Internal/External Rotation), Knee (Flexion/Extension), and Ankle (Dorsiflexion) divided by the normal range (American Academy of Orthopedic Surgeons and American Medical Association).
Time Frame: Baseline and at Week 105
Population: All participants for whom passive JROM were recorded at baseline and at Week 105.
Measure: Mean (Standard Error); unit: percentage of JROM
Arm/Group | Idursulfase (0.5 mg/kg, IV, Once-weekly)
Number analyzed (Participants) | 84
percentage of JROM | 0.63 (0.640)

3. Secondary Outcome: Change From Baseline in Mean Combined Liver and Spleen Volume at Week 105
Description: Determined by Magnetic Resonance Imaging (MRI). The change was calculated as Week 105 minus baseline.
Time Frame: Baseline and at Week 105
Population: All participants for whom combined liver and spleen volume were recorded at baseline and at Week 105.
Measure: Mean (Standard Error); unit: cubic centimeters (cc)
Arm/Group | Idursulfase (0.5 mg/kg, IV, Once-weekly)
Number analyzed (Participants) | 79
cubic centimeters (cc) | -325.5 (36.84)

4. Secondary Outcome: Change From Baseline in Mean Normalized Urine Glycosaminoglycans (GAG) Levels at Week 105
Description: Determined by urine testing. The change was calculated as Week 105 minus baseline.
Time Frame: Baseline and at Week 105
Population: All participants for whom normalized urine GAG levels were recorded at baseline and at Week 105.
Measure: Mean (Standard Error); unit: mcg GAG/mg creatinine
Arm/Group | Idursulfase (0.5 mg/kg, IV, Once-weekly)
Number analyzed (Participants) | 87
mcg GAG/mg creatinine | -238.25 (13.333)

5. Secondary Outcome: Change From Baseline in Mean Cardiac Left Ventricular Mass Index (LVMI) at Week 105
Description: Determined by echocardiogram. LVMI indexed to body surface area (g/m^2). The change was calculated as Week 105 minus baseline.
Time Frame: Baseline and at Week 105
Population: All participants for whom cardiac LVM were recorded at baseline and at Week 105.
Measure: Mean (Standard Error); unit: g/m^2
Arm/Group | Idursulfase (0.5 mg/kg, IV, Once-weekly)
Number analyzed (Participants) | 71
g/m^2 | 3.28 (3.826)

6. Primary Outcome: Change From Baseline in Mean Distance Walked in the 6-minute Walk Test (6MWT) at Week 105
Description: Determined on a walking course. The change was calculated as Week 105 minus baseline.
Time Frame: Baseline and at Week 105
Population: All participants for whom distance walked was recorded at baseline and at Week 105.
Measure: Mean (Standard Error); unit: meters (m)
Arm/Group | Idursulfase (0.5 mg/kg, IV, Once-weekly)
Number analyzed (Participants) | 85
meters (m) | 23.0 (7.94)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed throughout the duration of the TKT024EXT study. Adverse events were monitored from the time the first participant signed the informed consent until approximately 30 days after the last study visit.
Description: The "Serious Adverse Events" table lists all serious adverse events that occurred during the study regardless of a relationship to the study drug. The "Other Adverse Events" table lists those non-serious adverse events that were were determined to be possibly related to the study drug.
Arm/Group | Idursulfase (0.5 mg/kg, IV, Once-weekly)
Serious Adverse Events (participants affected / at risk) | 38/94
Other Adverse Events (participants affected / at risk) | 94/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idursulfase (0.5 mg/kg, IV, Once-weekly) (N=94)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1)
Abdominal Pain NOS (Gastrointestinal disorders) | 2 (2)
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 2 (2)
Acquired Claw Toe (Musculoskeletal and connective tissue disorders) | 1 (1)
Airway Complication of Anaesthesia (Injury, poisoning and procedural complications) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 2 (2)
Arrhythmia (Not Otherwise Specified [NOS]) (Cardiac disorders) | 1 (1)
Asthma Aggravated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) — 2 events of bacteraemia were at least possibly related to study drug as determined by the investigator.
Bronchopneumonia NOS (Infections and infestations) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 7 (7)
Catheter Related Complications (General disorders) | 1 (1)
Diarrhea NOS (Gastrointestinal disorders) | 1 (1)
Endocarditis Bacterial NOS (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Foreign Body Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hernia NOS (General disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Inguinal Hernia NOS (Gastrointestinal disorders) | 1 (1)
Joint Contracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Left Ventricular Failure (Cardiac disorders) | 1 (1)
Lobar Pneumonia NOS (Infections and infestations) | 1 (1)
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Obstructive Airways Disorder NOS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Otitis Media Chronic NOS (Infections and infestations) | 2 (2)
Otitis Media NOS (Infections and infestations) | 1 (1)
Otitis Media Serous Chronic NOS (Infections and infestations) | 1 (1)
Otitis Media Serous NOS (Infections and infestations) | 1 (1)
Pain in Foot (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericardial Effusions (Cardiac disorders) | 1 (1)
Pneumonia NOS (Infections and infestations) | 3 (3) — 1 event of pneumonia NOS was at least possibly related to study drug as determined by the investigator.
Poor Venous Access (Vascular disorders) | 10 (10) — 1 event of poor venous access was at least possibly related to study drug as determined by the investigator.
Psychosomatic Disease (Psychiatric disorders) | 1 (1)
Rash Macular (Skin and subcutaneous tissue disorders) | 1 (1) — This event of rash macular was at least possibly related to study drug as determined by the investigator.
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1)
Soft Tissue Infection NOS (Infections and infestations) | 1 (1)
Spinal Cord Compression NOS (Nervous system disorders) | 3 (4)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tympanic Membrane Disorder NOS (Ear and labyrinth disorders) | 1 (1)
Umbilical Hernia NOS (Gastrointestinal disorders) | 3 (3)
Upper Respiratory Tract Infection NOS (Infections and infestations) | 1 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Vomiting NOS (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idursulfase (0.5 mg/kg, IV, Once-weekly) (N=94)
Flushing (Vascular disorders) | 9 (32)
Hypotension NOS (Vascular disorders) | 6 (7)
Pallor (Vascular disorders) | 8 (8)
Seasonal allergy (Immune system disorders) | 6 (10)
Catheter site pain (General disorders) | 5 (5)
Chest pain (General disorders) | 9 (19)
Fall (General disorders) | 12 (19)
Fatigue (General disorders) | 12 (22)
Gait abnormal (General disorders) | 7 (8)
Influenza like illness (General disorders) | 11 (33)
Injection site extravasation (General disorders) | 6 (8)
Malaise (General disorders) | 7 (12)
Pain nos (General disorders) | 9 (16)
Pyrexia (General disorders) | 57 (187)
Rigors (General disorders) | 11 (17)
Abrasion nos (Injury, poisoning and procedural complications) | 17 (24)
Arthropod bite (Injury, poisoning and procedural complications) | 9 (11)
Head injury (Injury, poisoning and procedural complications) | 9 (9)
Limb injury nos (Injury, poisoning and procedural complications) | 7 (9)
Post procedural pain (Injury, poisoning and procedural complications) | 15 (25)
Thermal burn (Injury, poisoning and procedural complications) | 5 (6)
Neutrophil count decreased (Investigations) | 8 (8)
White blood cell count decreased (Investigations) | 5 (6)
Atrioventricular block first degree (Cardiac disorders) | 8 (9)
Dilatation atrial (Cardiac disorders) | 5 (6)
Tachycardia nos (Cardiac disorders) | 8 (24)
Ventricular hypertrophy (Cardiac disorders) | 6 (6)
Asthma nos (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Bronchitis nos (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Bronchospasm nos (Respiratory, thoracic and mediastinal disorders) | 8 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 53 (155)
Dyspnoea nos (Respiratory, thoracic and mediastinal disorders) | 14 (24)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (23)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 38 (100)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 39 (84)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 46 (102)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Rhinitis allergic nos (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Rhinitis nos (Respiratory, thoracic and mediastinal disorders) | 14 (20)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 31 (70)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 15 (28)
Anaemia nos (Blood and lymphatic system disorders) | 5 (5)
Carpal tunnel syndrome (Blood and lymphatic system disorders) | 19 (20)
Dizziness (Blood and lymphatic system disorders) | 18 (27)
Headache (Blood and lymphatic system disorders) | 53 (296)
Hypoaesthesia (Blood and lymphatic system disorders) | 8 (11)
Insomnia (Blood and lymphatic system disorders) | 5 (6)
Migraine nos (Blood and lymphatic system disorders) | 5 (6)
Conjunctivitis (Eye disorders) | 5 (5)
Visual acuity reduced (Eye disorders) | 5 (5)
Cerumen impaction (Ear and labyrinth disorders) | 13 (17)
Ear haemorrhage (Ear and labyrinth disorders) | 5 (5)
Ear pain (Ear and labyrinth disorders) | 24 (34)
Otorrhoea (Ear and labyrinth disorders) | 27 (88)
Abdominal pain nos (Gastrointestinal disorders) | 34 (73)
Constipation (Gastrointestinal disorders) | 11 (15)
Diarrhoea nos (Gastrointestinal disorders) | 32 (78)
Dyspepsia (Gastrointestinal disorders) | 7 (19)
Flatulence (Gastrointestinal disorders) | 5 (5)
Gastroenteritis nos (Gastrointestinal disorders) | 10 (12)
Loose stools (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 24 (44)
Toothache (Gastrointestinal disorders) | 7 (9)
Umbilical hernia nos (Gastrointestinal disorders) | 5 (5)
Vomiting nos (Gastrointestinal disorders) | 39 (102)
Hepatomegaly (Hepatobiliary disorders) | 5 (5)
Acne nos (Skin and subcutaneous tissue disorders) | 14 (17)
Contusion (Skin and subcutaneous tissue disorders) | 9 (10)
Eczema (Skin and subcutaneous tissue disorders) | 7 (9)
Erythema (Skin and subcutaneous tissue disorders) | 11 (35)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (27)
Rash macular (Skin and subcutaneous tissue disorders) | 6 (11)
Rash nos (Skin and subcutaneous tissue disorders) | 20 (60)
Rash papular (Skin and subcutaneous tissue disorders) | 6 (8)
Rash pruritic (Skin and subcutaneous tissue disorders) | 10 (16)
Skin lesion nos (Skin and subcutaneous tissue disorders) | 9 (13)
Urticaria nos (Skin and subcutaneous tissue disorders) | 14 (54)
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 (81)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (39)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 17 (24)
Pain in foot (Musculoskeletal and connective tissue disorders) | 5 (7)
Pain in limb (Musculoskeletal and connective tissue disorders) | 29 (59)
Ear infection nos (Infections and infestations) | 36 (91)
Furuncle (Infections and infestations) | 5 (5)
Influenza (Infections and infestations) | 7 (11)
Localised infection (Infections and infestations) | 5 (5)
Lower respiratory tract infection nos (Infections and infestations) | 7 (11)
Otitis media nos (Infections and infestations) | 22 (37)
Otitis media serous nos (Infections and infestations) | 7 (9)
Pneumonia nos (Infections and infestations) | 7 (9)
Respiratory tract infection nos (Infections and infestations) | 6 (12)
Sinusitis nos (Infections and infestations) | 9 (16)
Skin fungal infection nos (Infections and infestations) | 8 (9)
Tinea pedis (Infections and infestations) | 6 (21)
Tonsillitis (Infections and infestations) | 6 (6)
Tooth caries nos (Infections and infestations) | 7 (8)
Upper respiratory tract infection nos (Infections and infestations) | 47 (106)
Upper respiratory tract infection viral nos (Infections and infestations) | 9 (13)
Viral infection nos (Infections and infestations) | 10 (12)

LIMITATIONS AND CAVEATS:
This study design was open-label, and the lack of a concurrently followed placebo group limits the strength of the observations, because the progression of the disease is variable and has not been well described.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤ 180 days from the time submitted to Shire for review. Shire does not prohibit publication but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.